CLINICAL TRIAL: NCT04525430
Title: Comparison of Childbirth Education and Birth Plan With Childbirth Education Alone on Childbirth Self-Efficacy: A Randomized Controlled Trial
Brief Title: Childbirth Education and Birth Plan on Birth Self Efficacy in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, zeliha sunay, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/4-3
Record Dates: First submitted 2020-08-09; First posted 2020-08-25 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy Related; Self Efficacy
Keywords: pregnancy; childbirth education; birth plan; self efficacy; midwifery
MeSH Terms: interventions — Prenatal Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): only childbirth education group
  Interventions: Other: childbirth education
- Group 2 (Experimental): childbirth education and was subjected to a birth plan group
  Interventions: Other: childbirth education and was subjected to a birth plan
- Group 3 (No Intervention): standard care group

INTERVENTIONS:
Other: childbirth education — The 1st Session: General information about labor: Factors affecting labor, early signs of labor, signs of the start of labor, steps of labor, and procedures applied during labor.
  The 2nd Session: Methods of coping with birth contractions: Breathing exercises, relaxation exercises, massage, changing position, music, cold/warm application, focus, and walking.
  Other Names: group-ED
  Arms: Group 1
Other: childbirth education and was subjected to a birth plan — In the birth plan created by the researchers, the pregnant women considered the process from the start of labor to the end of labor and marked the expectation from and preferences about this process on the birth plan.
  Other Names: Group-ED&P
  Arms: Group 2

SUMMARY:
The pregnant women constituting the sample were divided into 3 groups. Group 1 was given only childbirth education (Group-ED), group 2 was given childbirth education and was subjected to a birth plan (Group-ED&P), and group 3 was the control group, each including 51 pregnant women.

DETAILED DESCRIPTION:
Aim: The purpose of this study was to investigate how pregnant women's childbirth self-efficacy was affected by childbirth education and birth plans applied with the education.

Methods: The research was carried out at seven Family Health Centers in Turkey as a randomized controlled trial. The pregnant women constituting the sample were divided into 3 groups. Group 1 was given only childbirth education (Group-ED), group 2 was given childbirth education and was subjected to a birth plan (Group-ED&P), and group 3 was the control group, each including 51 pregnant women.

ELIGIBILITY:
inclusion criteria:

* pregnant women who was in the third trimester (28-40 gestational weeks),
* who was literate or had a relative/helper who would write a birth plan to be prepared,
* who were not involved in any diagnosed risk at the present pregnancy (such as preeclampsia, diabetes, heart disease, placenta previa, oligohydramnios and multiple pregnancy)
* who did not have any diagnosed problems with the health of fetus (such as fetal anomaly and intrauterine growth retardation).

exclusion criteria:

• who had previous cesarean section were not included in the research.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change in birth self-efficacy level at 2 weeks (after intervention). | CBSEI was administered as a pretest to all pregnant women in the three groups. After two weeks CBSEI was administered as a posttest to the pregnant women in all three groups.
  Childbirth Self-Efficacy was measured with Childbirth Self-Efficacy Inventory (CBSEI) Short Version. The scale consisted of two sub-dimensions, self-efficacy expectancy and outcome expectancy. The highest score to be taken from the sub-dimensions was 160, and the lowest score was 16. Pregnant women's having a high score on this scale meant that the level of their childbirth self-efficacy was high.

CONTACTS AND LOCATIONS:
Overall Officials: zeliha sunay, Msc, Principal Investigator — munzur üniversitesi
Locations (1):
- İnönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Result] Aragon M, Chhoa E, Dayan R, Kluftinger A, Lohn Z, Buhler K. Perspectives of expectant women and health care providers on birth plans. J Obstet Gynaecol Can. 2013 Nov;35(11):979-985. doi: 10.1016/S1701-2163(15)30785-4. PMID 24246397
- See also: citation link — https://pubmed.ncbi.nlm.nih.gov/24246397/